CLINICAL TRIAL: NCT05852067
Title: The Second Affiliated Hospital Zhejiang University School od Medicine
Brief Title: Effects of Prolonged Continuous Theta Burst Stimulation on Pain and Neural Excitability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2023-0276
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: pcTBS; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation of M1 (Experimental): pcTBS was administered to the left M1 at 80% resting motor threshold (RMT), consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz. A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline.
  Interventions: Device: pcTBS of M1
- SHAM stimulation (Sham Comparator): The Sham stimulation was delivered using the same protocol, with the coil being orientated at 90° to the scalp so that the magnetic field would be delivered away from the scal
  Interventions: Device: SHAM stimulation

INTERVENTIONS:
Device: pcTBS of M1 — Prolonged continuous theta-burst stimulation (pcTBS) was administered to the left M1 at 80% RMT, consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz. A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline
  Arms: Active stimulation of M1
Device: SHAM stimulation — The Sham stimulation was delivered using the same pcTBS protocol, with the coil being flipped 90◦to the scalp so that the magnetic field would be delivered away from the scalp
  Arms: SHAM stimulation

SUMMARY:
Numerous studies have confirmed the analgesic effect of M1-rTMS on both induced pain and various chronic pains and subsequently found that pcTBS is more time-efficient and can produce the same or even stronger analgesic effect, however, its study in pathological pain h has not been thoroughly investigated. Due to the dynamic nature of the injury sensory system, pain also exhibits a dynamic process, but there is a lack of specific methods or biomarkers to document this process. Surface electromyography (EMG) is a common technique used in rTMS studies to reflect changes in cortical excitability. In turn, both pain and rTMS interventions can cause changes and thus can be used as a potential biomarker to predict pain onset and progression. In addition, the number of sessions of rTMS treatment is an important factor influencing the analgesic effect of rTMS. In summary, this study intends to explore the best pain predictor by using a capsaicin-induced pain model in healthy volunteers, monitor the dynamic changes of cortical excitability index and VAS score before and after pcTBS intervention, and also verify the relationship between the number of pcTBS treatments and analgesic effect, to provide a new strategy for the prevention and treatment of neuropathic pain.

DETAILED DESCRIPTION:
This study was a prospective, single-blind, sham-controlled, crossover-design trial. Each subject was randomized to receive 3 sessions of rTMS intervention, consisting of 2 consecutive pcTBS stimulations and 1 sham stimulation, with no less than 3 days between each session. The pain was induced by applying capsaicin to the dorsum t of the right hand and recording electromyographic (EMG) signals with surface electrodes on the right first interosseous muscle. Subjects received M1- pcTBS or sham stimulation (Sham) intervention at 40 minutes of capsaicin application (T40). Subjects' cortical excitability was measured at 5-minute intervals at baseline, 40 minutes after capsaicin application and pcTBS intervention, and pain perception was assessed at 10-minute intervals (each assessment to be performed at the end of the measurement).

ELIGIBILITY:
Inclusion Criteria:

1) 18-65 years of age; 2) physical and mental health, free of chronic pain (through interviews and McGill questionnaires); 3) Right-handed

Exclusion Criteria:

1) inability to receive TMS interventions (e.g. pacemaker); 2) mental illness or suicidal tendencies; 3) history of previous seizures/epilepsy; 4) previous craniocerebral surgery for stroke or other reasons; 5) drug/substance dependence; 6) Inability to sit upright to cooperate with assessment and treatment; 7) Pregnancy or planning to become pregnant within half a year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
change of pain intensity | through study completion, an average of 6 months
  pain intensity on a 10-cm visual analogue scale (VAS) extending from 0 (no pain) to 100 (maximal pain possible) at baseline and posttreatment of pcTBS stimulation

SECONDARY OUTCOMES:
Motor-evoked potential (MEP) | through study completion, an average of 6 months
  Corticospinal excitability was measured with MEP at rest of the first dorsal interosseous (FDI) muscle, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward)
Cortical silent period (CSP) | through study completion, an average of 6 months
  Corticospinal excitability will be measured with CSP during a sustained voluntary FDI muscle contraction, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward)
pain intensity after two sessions of pcTBS | through study completion, an average of 6 months
  pain intensity on a 10-cm visual analogue scale (VAS) extending from 0 (no pain) to 100 (maximal pain possible) after two sessions of pcTBS

CONTACTS AND LOCATIONS:
Overall Officials: min yan, prof., Study Chair — The second affiliated hospital of Zhejiang University hangzhou
Locations (1):
- The second affiliated hospital of Zhejiang University hangzhou, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No